CLINICAL TRIAL: NCT06571604
Title: Preoperative Gluteal Muscle Atrophy: A Silent Predictor of THA Dislocation.
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: THAdislocation glutealatrophy
Record Dates: First submitted 2024-08-23; First posted 2024-08-26 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-08

CONDITIONS: Dislocation; Total Hip Arthroplasty; Muscle Degeneration
Keywords: Total Hip Arthroplasty; Muscle Fatty Degeneration; CT; Gluteal Muscles
MeSH Terms: conditions — Joint Dislocations

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Dislocation group: Patients who underwent primary total hip arthroplasty with preoperative CT-scan and encountered an episode of dislocation.
  Interventions: Diagnostic Test: Dislocation
- Control group: Patients underwent primary total hip arthroplasty with preoperative CT-scan, who did not experience any episodes of dislocation within two years post-surgery, adhering to the previously outlined exclusion criteria (group control).
  Interventions: Diagnostic Test: No dislocation

INTERVENTIONS:
Diagnostic Test: Dislocation — One episode of total hip dislocation diagnozied on Xray within 2 years of surgery
  Groups: Dislocation group
Diagnostic Test: No dislocation — No experience of dislocation within two years post-surgery
  Groups: Control group

SUMMARY:
This study looks at how fat buildup in hip muscles relates to hip osteoarthritis and less favorable recovery after hip replacement surgery. While it is known that weak gluteal muscles might cause problems, it is not yet proven if this specifically leads to hip dislocation after surgery. The goal of this study is to compare fat buildup in gluteal muscles between patients who had a hip dislocation soon after surgery and those who did not.

ELIGIBILITY:
Inclusion Criteria:

* primary THA with preoperative CT-scan

Exclusion Criteria:

* malposition of acetabular implants outside the Lewinneck safe zone,
* neurological or cognitive disorders,
* associated spinal pathologies (within the context of a hip-spine syndrome),
* chronic alcoholism,
* aseptic osteonecrosis,
* revision surgeries,
* late dislocations attributed to polyethylene wear,
* replacement following post-traumatic coxarthrosis due to acetabulum injuries.
* diameters of the prosthetic heads ≠ 32mm

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients following THA at Nimes university hospital
Sampling Method: Non-Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2023-05-01 (Actual)

PRIMARY OUTCOMES:
Mean Attenuation Ratio | The CT scan of the pelvis used to plan the operation is performed between one and two months before the surgery.
  The mean attenuation ratio (MAR), representing muscle fat degeneration, corresponds to the mean grayscale pixels in the selected area, expressed in Hounsfield Units (HU). Subsequently, the segmentation process was applied, selectively retaining pixels within the range of -30 HU to 150 HU. This range corresponds to muscle fibers and intramuscular fat, effectively excluding extra-fascial fat and bone pixels.

SECONDARY OUTCOMES:
Cross-Sectional Area | The CT scan of the pelvis used to plan the operation is performed between one and two months before the surgery.
  The cross-sectional area (CSA), measured in square centimeters (cm²) defines the average muscle surface area.
Intramuscular Fatty Fraction | The CT scan of the pelvis used to plan the operation is performed between one and two months before the surgery.
  Finally, the intramuscular fatty fraction (IFF) or percentage of intramuscular fat was calculated using the IB Delta Suite plug-in with thresholds of -30/0/150. Pixels below -30 HU and above 150 HU were designated as extra-muscular, while pixels ranging between 0 HU and 150 HU represented muscle fibers. Pixels falling between -30 HU and 0 HU denoted intramuscular fat, constituting the IFF.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Nîmes, Nîmes, Gard, France